CLINICAL TRIAL: NCT02127099
Title: The Incidence of Undiagnosed OSA in Multi-ethic Races of Malaysia and the Associated Postoperative Complications
Brief Title: The Incidence of Undiagnosed OSA Compared in Multi-ethic Races of Malaysia & the Associated Postoperative Complications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Wang Chew Yin, Professor, University of Malaya
Other Study IDs: 1017.8
Record Dates: First submitted 2014-04-25; First posted 2014-04-30 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; obstructive; sleep; apnea; operation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with OSA: Post operative patients with OSA
- Post-operative Patients without OSA: All post operative patients without OSA

SUMMARY:
Obstructive sleep apnoea (OSA) is a condition in which a person's sleep is disrupted with momentary periods of apnoea and hypopnoea. This occurs when there is a blockage to airflow. When this happens, the patient will snore, gasp or choke in the attempt to attain more oxygen. This results in disrupted sleep and the patient may even awake from sleep.

It has been found that a great proportion of Malaysians have habitual snoring and with the increase in obesity over the years, it is a concern that OSA may be prevalent in Malaysia.

However, it has been seen that OSA is commonly undiagnosed in patient. This poses a worry because these people can come in for surgery. Diagnosis of OSA before surgery is important in order to prepare for the complication related to OSA.

DETAILED DESCRIPTION:
Research staff will interview and examine patients and review their charts to obtain information on patient characteristics. Patients will also be assessed using STOP-BANG Questionnaire & Epworth Sleepiness Scale.

Anaesthesia and surgery will be performed according to routine standard of care.

Drugs used during anaesthesia, postoperative analgesia and hemodynamic data will be recorded.

During their stay in hospital, patients will be followed daily, and outcomes will be recorded, until discharge. Data on medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult males and females
* age ≥ 18 years
* undergoing elective surgery ( general,regional or local anaesthesia with monitored anaesthesia care)

Exclusion Criteria:

* previous diagnosis of OSA or any sleep-related breathing disorder
* they are unwilling
* their surgery included tonsillectomy, septoplasty, uvloplasty, pharyngoplasty, tracheostomy, or prolonged mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients over age 18 undergoing non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of OSA | 30 days
  Incidence of OSA in surgical patients among the ethnic races.

SECONDARY OUTCOMES:
Post-operative complications | 30 days
  Any cardiovascular or respiratory complications detected during the post-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Chew Yin Wang, MBChB, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia